CLINICAL TRIAL: NCT03121430
Title: The Safety and Efficacy of Drug Eluting Peripheral Vascular Stent System for the Treatment of Superficial Femoral Artery Stenosis and /or Occlusion: a Multi-center Stratified Randomized Single- Blind Controlled Trial
Brief Title: Study of Drug Eluting Peripheral Vascular Stent System in Superficial Femoral Artery Stenosis and /or Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Zylox Medical Device Co., Ltd. (Industry)
Collaborators: Guangzhou Osmunda Medical Device Technology, Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2052108140
Record Dates: First submitted 2017-04-09; First posted 2017-04-20 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Disease; Superficial Femoral Artery Stenosis; Superficial Femoral Artery Occlusion
Keywords: peripheral arterial disease; Drug eluting peripheral vascular stent system; primary patency
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): subjects using the drug eluting peripheral vascular stent system
  Interventions: Device: Drug eluting peripheral vascular stent system
- Group B (Active Comparator): subjects using the Nitinol Stent System (Cordis Corporation)
  Interventions: Device: Nitinol Stent System

INTERVENTIONS:
Device: Drug eluting peripheral vascular stent system — Drug eluting peripheral vascular stent system、Color Doppler Ultrasonography (CDU) imaging、Dual Fluoroscopic Imaging、Digital subtraction angiography（DSA）
  Arms: Group A
Device: Nitinol Stent System — Nitinol Stent System、Color Doppler Ultrasonography (CDU) imaging and Dual Fluoroscopic Imaging、Digital subtraction angiography（DSA）
  Other Names: Cordis Corporation
  Arms: Group B

SUMMARY:
Evaluation of drug eluting peripheral vascular stent system for the treatment of superficial femoral artery stenosis and / or occlusion, there is better in effectiveness and clinical performance compared with similar products already on the market.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized study designed to enroll 138 patients with superficial femoral artery stenosis and /or occlusion who will be randomized 1:1 to be treated with the Drug eluting peripheral vascular stent system versus the commercially available Nitinol Stent System (Cordis Corporation). Patients will receive Color Doppler Ultrasonography (CDU) imaging and Dual Fluoroscopic Imaging at 6th month and 12th month post procedure. Clinical visits are scheduled at 0~30 days, 6 months, 12 months, and telephone visits are scheduled at 1 month, 3months, and 9 months. Furthermore, CDU will also be performed at baseline in all participants of the study.

ELIGIBILITY:
Inclusion Criteria in Preoperative:

* Aged from 18 to 85 years old, male or female
* Subject's target lesions were stenosis and/or occlusion
* Subject is aware of the study content, showing sufficient compliance with the research protocol and sign the Informed Consent

Exclusion Criteria in Preoperative:

* In-Stent Restenosis(IRS) or restenosis after drug-eluting balloon administration
* Serum creatinine concentration of the subject is higher than 1.5 times of the upper limit of normal serum creatinine concentration
* Subject with coagulation abnormalities should not be performed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
primary patency rate at 12 months after operation | 12 months
  the rate of the target lesion diameter stenosis <50% patients confirmed by Color Doppler Ultrasonography (CDU) imaging at 12 months postoperatively

SECONDARY OUTCOMES:
primary patency rate at 6 months after operation | 6 months
  the rate of the target lesion diameter stenosis <50% patients confirmed by Color Doppler Ultrasonography (CDU) imaging at 6 months postoperatively
target lesion revascularization rate | Preoperative，up to 1 month，6 months，12 months
  subject found that the presence of restenosis in the target lesion in follow-up , and need to re-intervention or bypass graft according to the clinical symptoms
Stent fracture rate | 6 months、12 months
  using the Dual Fluoroscopic Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhong, Principal Investigator — Beijing Anzhen Hospital; Guo Wei, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, China

IPD SHARING:
Plan to Share IPD: No